CLINICAL TRIAL: NCT01811264
Title: Improving Psychosocial Quality of Life in Women With Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Marla L Clayman, Adjunct Faculty, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PPA Study
Record Dates: First submitted 2013-02-19; First posted 2013-03-14 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: Metastatic; Quality of life; Decision making
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will begin with a pre-visit structured interview to determine emotional and physical well-being, anxiety, depression, and self-efficacy. Then they will be helped through the Patient-Participation Aid (PPA) by the research assistant (RA). Then they will meet with their doctor while the visit is video-recorded. After they will complete a post-visit interview to see if there were any health decisions made, patients level of involvement, and doctor communication. Follow up phone interviews will be conducted at 1 week and 3 months to assess patients self-reported changes in well-being, anxiety, depression, and decision regret.
  Interventions: Behavioral: Patient-Participation Aid
- Usual Care (No Intervention): Participants will begin with a pre-visit structured interview to determine emotional and physical well-being, anxiety, depression, and self-efficacy. They will have their doctor's visit video recorded. After they will complete a post-visit interview to see if there were any health decisions made, patients level of involvement, and doctor communication.Follow up phone interviews will be conducted at 1 week and 3 months to assess patients self-reported changes in well-being, anxiety, depression, and decision regret.

INTERVENTIONS:
Behavioral: Patient-Participation Aid — The PPA consists of a folder that addresses the three behaviors we hope to influence: agenda setting, asking questions, and making preferences known. The information inside contains sample questions for each section, with room for the patient to write her own questions. Each section models behavior by giving context for the items and specific example questions. It also addresses barriers to understanding by indicating that it is acceptable to ask questions when something is not clear or terms are unfamiliar.
  Other Names: PPA
  Arms: Intervention

SUMMARY:
Through a patient participation aid (PPA) the investigators hope to improve the psychosocial well-being of women diagnosed with metastatic breast cancer by empowering them to be active participants in clinical encounters.

DETAILED DESCRIPTION:
The team has developed a brief Patient Participation Aid (PPA) to promote patient health literacy and encourage women to be active in the decisions that are being made about their healthcare which will lead to their satisfaction with healthcare and improves their psychosocial well-being. The paper-based PPA uses adult learning principles to limit and sequence plain language messages that have been framed from a patient's perspective. The PPA uses theory-based design to increase patients' involvement in the medical visit by modeling - through text and images - how a patient can: 1) set the visit agenda, 2) formulate questions, and 3) assert personal preferences. The specific aims of this study are to: 1- Assess the effectiveness of the PPA to increase patient involvement during clinical encounters. 2- Evaluate the effectiveness of the PPA to improve patient psychosocial outcomes. 3- Explore if the effect of the PPA varies by patients' literacy skills. To achieve this aims, the investigators will conduct a randomized controlled trial to evaluate the PPA among patients with a new diagnosis or progression of metastatic breast cancer at two cancer centers that serve diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

* female patients with metastatic breast cancer seeing one of the study physicians at one of the identified study clinics
* age 21 or older
* having suspected progression of metastatic disease

Exclusion Criteria:

* patients with an uncorrectable hearing impairment or having limited English proficiency, as this would adversely affect their ability to communicate with the physician
* patients with uncorrectable vision impairment, as this would make it impractical for the patient to read the intervention
* patients too ill to meaningfully converse with the physician

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-12; Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - General (FACT-G) | Change in functional assessment of cancer therapy from pre-visit at 3 months post-visit
  Evaluated at 30 minutes prior to, one week after, and 3 months after the patients visit with their doctor, this measure collects scales of the social and family well-being, emotional well-being, and functional well-being.

SECONDARY OUTCOMES:
Rapid Estimate of Adult Literacy in Medicine (REALM-SF) | Pre-Visit
  A 7-item word recognition test to provide clinicians with a valid quick assessment of patient health literacy.

OTHER OUTCOMES:
Decision Regret Scale | Change in decision regret from pre-visit at 3 months post-visit
  Collected at post-visit, and follow-ups, this measures the patient's regret and feelings regarding the most recent treatment-related decision

CONTACTS AND LOCATIONS:
Overall Officials: Marla Clayman, Ph.D, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - H Lee Moffitt Comprehensive Cancer Center, Tampa, Florida
  - Feist-Weiller Cancer Center, Shreveport, Louisiana

IPD SHARING:
Plan to Share IPD: No